CLINICAL TRIAL: NCT01316913
Title: A Multi-center Trial Comparing the Efficacy and Safety of GSK573719/GW642444 With GSK573719 and With Tiotropium Over 24 Weeks in Subjects With COPD
Brief Title: 24-week Trial Comparing GSK573719/GW642444 With GSK573719 and With Tiotropium in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113374
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: tiotropium; long-acting muscarinic antagonist; COPD; long-acting beta agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK573719/GW642444 125/25 (Experimental): 125/25 mcg once-daily
  Interventions: Drug: GSK573719/GW642444 125/25
- GSK573719/GW642444 62.5/25 (Experimental): 62.5/25 mcg once-daily
  Interventions: Drug: GSK573719/GW642444 62.5/25
- GSK573719 (Experimental): 125 mcg once-daily
  Interventions: Drug: GSK573719
- tiotropium bromide (Active Comparator): 18 mcg once-daily
  Interventions: Drug: tiotropium bromide

INTERVENTIONS:
Drug: GSK573719/GW642444 125/25 — 125/25 mcg once-daily
  Other Names: GSK573719/vilanterol trifenatate
  Arms: GSK573719/GW642444 125/25
Drug: GSK573719/GW642444 62.5/25 — 62.5/25 mcg once-daily
  Other Names: GSK573719/vilanterol trifenatate
  Arms: GSK573719/GW642444 62.5/25
Drug: GSK573719 — 125 mcg once-daily
  Arms: GSK573719
Drug: tiotropium bromide — 18 mcg once-daily
  Arms: tiotropium bromide

SUMMARY:
This is a Phase III multicenter, randomized, double-blind, double-dummy, parallel-group study to evaluate the efficacy and safety of two doses of GSK573719/GW642444 Inhalation Powder, GSK573719 Inhalation Powder via a Novel Dry Powder Inhaler and tiotropium via HandiHaler when administered once-daily over a 24-week treatment period in subjects with chronic obstructive pulmonary disease (COPD). Subjects who meet eligibility criteria at Screening (Visit 1) will complete a 7 to10 day run-in period followed by a randomization visit (Visit 2) then a 24-week treatment period. There will be a total of 9 clinic study visits. A follow-up phone contact for adverse event assessment will be conducted approximately one week after the last study visit (Visit 9 or Early Withdrawal). The total duration of subject participation in the study will be approximately 26 weeks. The primary measure of efficacy is clinic visit trough (pre-bronchodilator and pre-dose) forced expiratory volume in one second (FEV1) on Treatment Day 169. Safety will be assessed by adverse events, 12-lead ECGs, vital signs, and clinical laboratory tests.

DETAILED DESCRIPTION:
This is a 24-week, Phase III multicenter, randomized, double-blind, double-dummy, parallel-group study. Eligible subjects will be randomized to GSK573719/GW642444 125/25mcg, GSK573719/GW642444 62.5/25mcg, GSK573719 125mcg, or tiotropium treatment groups in a 1:1:1:1 ratio. Treatments will be administered once-daily in the morning by inhalation using a Novel Dry Powder Inhaler (Novel DPI) and HandiHaler. There will be a total of 9 study clinic visits conducted on an outpatient basis. Subjects who meet the eligibility criteria at Screening (Visit 1) will complete a 7 to 10 day run-in period followed by a 24-week treatment period. Clinic visits will be at Screening, Randomization (Day 1), Day 2, after 4, 8, 12, 16, and 24-weeks of treatment, and 1 day after the Week 24 Visit (also referred as Treatment Day 169). A follow-up contact for adverse assessment will be conducted by telephone approximately 7 days after Visit 9 or the Early Withdrawal Visit. The total duration of subject participation, including follow-up will be approximately 26 weeks. All subjects will be provided with albuterol/salbutamol for use on an "as-needed" basis throughout the run-in and study treatment periods. At screening, pre-bronchodilator spirometry testing will be followed by post-albuterol/salbutamol spirometry testing. Post-albuterol/salbutamol FEV1 and FEV1/forced vital capacity (FVC) values will be used to determine subject eligibility. To further characterize bronchodilator responsiveness, post-ipratropium testing will be conducted following completion of post-albuterol/salbutamol spirometry. Spirometry will be conducted at each post-randomization clinic visit. Six hour post-dose serial spirometry will be conducted at Visits 2, 6, and 8. Trough spirometry will be obtained 23 and 24 hours after the previous day's dose of blinded study medication at Visits 3 to 9. All subjects will be provided with an electronic diary (eDiary) for completion daily in the morning and the evening throughout the run-in and treatment periods. Subjects will use the eDiary to record peak expiratory flow (PEF) each morning, dyspnea scores using the Shortness of Breath with Daily Activities instrument (SOBDA), daily use of supplemental albuterol/salbutamol as either puffs/day from a metered-dose inhaler (MDI) and/or nebules used per day, and any healthcare contacts related to COPD. Additional assessments of dyspnea will be obtained using the Baseline and Transition Dyspnea Index (BDI/TDI) which is an interviewer based instrument. At Visit 2, the severity of dyspnea at baseline will be assessed using the BDI. At subsequent visits (Visits 4, 6, and 8) change from baseline will be assessed using the TDI. General health status will be evaluated using the subject-completed EQ-5D questionnaire at Visits 2, 4, 6, and 8. Disease specific health status will be evaluated using the subject-completed St. George's Respiratory Questionnaire (SGRQ) at Visits 2, 4, 6, and 8, and the subject-completed COPD Assessment Test (CAT) at Visits 2, 6, and 8. The occurrence of adverse events will be evaluated throughout the study beginning at Visit 2. SAEs will be collected over the same time period as for AEs. However, any SAEs assessed as related to study participation (e.g., study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK concomitant medication, will be recorded from the time a subject consents to participate in the study up to and including any follow up contact. Additional safety assessments of vital signs (blood pressure and pulse rate), 12-lead ECGs and standard clinical laboratory tests (hematology and chemistry) will be obtained at selected clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* outpatient
* signed and dated written informed consent
* 40 years of age or older
* male and female subjects
* COPD diagnosis
* at least 10 pack-year smoking history
* post-albuterol/salbutamol FEV1/FVC ratio of <0.70 and post-albuterol/salbutamol FEV1 of less than or equal to 70% predicted normal values
* score of greater than or equal to 2 on the Modified Medical Resarch Council Dyspnea Scale (mMRC)

Exclusion Criteria:

* women who are pregnant or lactating or are planning on becoming pregnant during the study
* current diagnosis of asthma
* other respiratory disorders other than COPD
* other diseases/abnormalities that are uncontrolled including cancer not in remission for at least 5 years
* chest x-ray or CT scan with clinically significant abnormalities not believed to be due to COPD
* hypersensitivity to anticholinergics, beta-agonists, lactose/milk protein or magnesium stearate or medical conditions associated with inhaled anticholinergics
* hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1
* lung volume reduction surgery within 12 months prior to Visit 1
* abnormal and clinically significant ECG at Visit 1
* significantly abnormal finding from laboratory tests at Visit 1
* unable to withhold albuterol/salbutamol at least 4 hours prior to spirometry at each visit
* use of depot corticosteroids within 12 weeks of Visit 1
* use of oral or parenteral corticosteroids, antibiotics for lower respiratory tract infection, or cytochrome P450 3A4 inhibitors, within 6 weeks of Visit 1
* use of long-acting beta-agonist (LABA)/inhaled corticosteroid (ICS) product if LABA/ICS therapy is discontinued withing 30 days of Visit 1
* use of ICS at a dose of >1000mcg/day of fluticasone propionate or equivalent within 30 days of Visit 1
* initiation or discontinuation of ICS within 30 days of Visit 1
* use of tiotropium or roflumilast within 14 days of Visit 1
* use of theophyllines, oral leukotriene inhibitors, long-acting oral beta-agonists, or inhaled long-acting beta-agonists within 48 hours of Visit 1
* short-acting oral beta-agonists within 12 hours of Visit 1
* use of LABA/ICS combination products only if discontinuing LABA therapy and switching to ICS monotherapy within 48 hours of Visit 1 for the LABA component
* use of sodium cromoglycate or nedocromil sodium within 24 hours of Visit 1
* use of inhaled short-acting beta-agonists, inhaled short-acting anticholinergics, or inhaled short-acting anticholinergic/short-acting beta-agonist combination products within 4 hours of Visit 1
* use of any other investigational medication within 30 days or 5 drug half-lives (whichever is longer)
* long-term oxygen therapy prescribed for >12 hours per day
* regular use of nebulized short-acting bronchodilators
* participation in acute phase of pulmonary rehabilitation program
* known or suspected history of alcohol or drug abse within 2 years prior to Visit 1
* anyone affiliated with the investigator site (e.g., investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member)
* previous exposure to GSK573719, GSK573719/GW642444 combination, GW642444 (vilanterol), or fluticasone furoate/GW642444 combination

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 872 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (84):
- United States (20):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Morgantown, West Virginia
- Argentina (4):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Mendoza, Mendoza Province
  - GSK Investigational Site, Buenos Aires
- Australia (9):
  - GSK Investigational Site, Concord, New South Wales
  - GSK Investigational Site, Cairns, Queensland
  - GSK Investigational Site, Carina Heights, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Daw Park, South Australia
  - GSK Investigational Site, Frankston, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (9):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, St-Romulad, Quebec
- Chile (4):
  - GSK Investigational Site, Port Montt, Los Lagos Region
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Talca, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Germany (15):
  - GSK Investigational Site, Schwetzingen, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Oranienburg, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Schwedt, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- Mexico (4):
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México
- Romania (3):
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Târgovişte
- South Africa (8):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Boksburg North
  - GSK Investigational Site, Die Wilgers
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Groenkloof
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Thabazimbi
- South Korea (8):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seongnam-si, Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Maleki-Yazdi MR, Singh D, Anzueto A, Tombs L, Fahy WA, Naya I. Assessing Short-term Deterioration in Maintenance-naive Patients with COPD Receiving Umeclidinium/Vilanterol and Tiotropium: A Pooled Analysis of Three Randomized Trials. Adv Ther. 2017 Jan;33(12):2188-2199. doi: 10.1007/s12325-016-0430-6. Epub 2016 Oct 28. PMID 27796912
- [Derived] Decramer M, Anzueto A, Kerwin E, Kaelin T, Richard N, Crater G, Tabberer M, Harris S, Church A. Efficacy and safety of umeclidinium plus vilanterol versus tiotropium, vilanterol, or umeclidinium monotherapies over 24 weeks in patients with chronic obstructive pulmonary disease: results from two multicentre, blinded, randomised controlled trials. Lancet Respir Med. 2014 Jun;2(6):472-86. doi: 10.1016/S2213-2600(14)70065-7. Epub 2014 May 14. PMID 24835833
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113374 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113374 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113374 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113374 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113374 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113374 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113374 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria at Screening (Visit 1) completed a 7- to10-day run-in period and were then randomized to a 24-week treatment period. A total of 1191 par. were screened; 872 par. were randomized and 869 par. entered the treatment period.
Groups:
- UMEC 125 µg QD: Participants received umeclidinium bromide (UMEC) 125 micrograms (µg) once daily (QD) via a dry powder inhaler (DPI) and placebo QD via a HandiHaler in the morning for 24 weeks.
- UMEC/VI 62.5/25 µg QD: Participants received umeclidinium bromide/vilanterol (UMEC/VI) 62.5/25 µg QD via a DPI and placebo QD via a HandiHaler in the morning for 24 weeks.
- UMEC/VI 125/25 µg QD: Participants received UMEC/VI 125/25 µg QD via a DPI and placebo QD via a HandiHaler in the morning for 24 weeks.
- TIO18 µg QD: Participants received tiotropium bromide (TIO) 18 µg QD via a HandiHaler and placebo QD via a DPI in the morning for 24 weeks.
Period: Overall Study
Arm/Group | UMEC 125 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD | TIO18 µg QD
Started | 222 | 217 | 215 | 215
Completed | 165 | 163 | 166 | 176
Not Completed | 57 | 54 | 49 | 39
Not completed — Adverse Event | 17 | 20 | 15 | 11
Not completed — Lack of Efficacy | 22 | 12 | 9 | 13
Not completed — Protocol Violation | 1 | 4 | 4 | 1
Not completed — Protocol-defined Stopping Criteria | 7 | 8 | 11 | 6
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 10 | 9 | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- UMEC 125 µg QD: Participants received UMEC 125 µg QD via a DPI and placebo QD via a HandiHaler in the morning for 24 weeks.
- UMEC/VI 62.5/25 µg QD: Participants received UMEC/VI 62.5/25 µg QD via a DPI and placebo QD via a HandiHaler in the morning for 24 weeks.
- TIO18 µg QD: Participants received TIO 18 µg QD via a HandiHaler and placebo QD via a DPI in the morning for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | UMEC 125 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD | TIO18 µg QD | Total
Number analyzed (Participants) | 222 | 217 | 215 | 215 | 869
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (8.33) | 65.0 (8.62) | 63.8 (8.51) | 65.2 (8.30) | 64.6 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 77 | 67 | 62 | 280
  Male | 148 | 140 | 148 | 153 | 589
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 6 | 8 | 9 | 8 | 31
  Asian - East Asian Heritage | 35 | 34 | 36 | 34 | 139
  Asian - South East Asian Heritage | 2 | 1 | 1 | 2 | 6
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 0 | 1
  White - Arabic/North African Heritage | 1 | 0 | 0 | 0 | 1
  White - White/Caucasian/European Heritage | 169 | 163 | 160 | 163 | 655
  White - Mixed Race | 0 | 1 | 0 | 0 | 1
  Mixed Race | 9 | 9 | 9 | 8 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinic Visit Trough Forced Expiratory Volume in One Second (FEV1) at Day 169
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 measurements were taken electronically by spirometry on Days 2, 28, 56, 84, 112, 168, and 169. Baseline is defined as the mean of the assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1. Trough FEV1 is defined as the mean of the FEV1 values obtained at 23 and 24 hours after the previous morning's dosing (i.e., trough FEV1 on Day 169 is the mean of the FEV1 values obtained 23 and 24 hours after the morning dosing on Day 168). Change from Baseline at a particular visit was calculated as the trough FEV1 at that visit minus Baseline. Analysis was performed using a repeated measures model with covariates of treatment, Baseline, smoking status, center group, day, and day by Baseline and day by treatment interactions. ITT=Intent-to-Treat.
Time Frame: Baseline and Day 169
Population: ITT Population: all participants randomized to treatment who received at least one dose of randomized study drug in the Treatment Period. Participants analyzed are those with data available at the presented time point; but, all participants without missing covariate information and with >=1 post-Baseline measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- UMEC/VI 125/25 QD: Participants received UMEC/VI 125/25 µg QD via a DPI and placebo QD via a HandiHaler in the morning for 24 weeks.
Arm/Group | UMEC 125 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 QD | TIO18 µg QD
Number analyzed (Participants) | 163 | 161 | 164 | 175
Liters | 0.186 (0.0178) | 0.208 (0.0180) | 0.223 (0.0179) | 0.149 (0.0176)
Statistical Analysis 1: Comparison: UMEC 125 µg QD vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p = 0.377, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.022, 95% CI 2-sided [-0.027 to 0.072] — Least squares mean difference=UMEC/VI 62.5/25 µg minus UMEC 125 µg
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 µg QD vs TIO18 µg QD; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis — nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.060, 95% CI 2-sided [0.010 to 0.109] — Least squares mean difference=UMEC/VI 62.5/25 µg minus TIO 18 µg
Statistical Analysis 3: Comparison: UMEC 125 µg QD vs UMEC/VI 125/25 QD; Test type: Superiority or Other; p = 0.142, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.037, 95% CI 2-sided [-0.012 to 0.087] — Least squares mean difference=UMEC/VI 125/25 µg minus UMEC 125 µg
Statistical Analysis 4: Comparison: UMEC/VI 125/25 QD vs TIO18 µg QD; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.074, 95% CI 2-sided [0.025 to 0.123] — Least squares mean difference=UMEC/VI 125/25 µg minus TIO 18 µg

2. Secondary Outcome: Change From Baseline (BL) in Weighted Mean (WM) 0-6 Hour FEV1 Obtained Post-dose at Day 168
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The WM FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The WM was calculated at Days 1, 84, and Day 168 using the 0-6-hour post-dose FEV1 measurements collected on that day, which included pre-dose (Day 1: 30 minutes [min] and 5 min prior to dosing; other serial visits: 23 and 24 hours after the previous morning dose) and post-dose at 15 minutes, 30 minutes, 1 hour, 3 hours, and 6 hours. Change from BL at a particular visit was calculated as WM at that visit minus BL. Analysis was performed using a repeated measures model with covariates of treatment, BL (mean of the two assessments made 30 minutes and 5 minutes pre-dose on Day 1), smoking status, center group, day, and day by BL and day by treatment interactions.
Time Frame: Baseline and Day 168
Population: ITT Population. Par. analyzed are those with data available at the presented time point; but, all par. without missing covariate information and with >=1 post-Baseline measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC 125 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD | TIO18 µg QD
Number analyzed (Participants) | 161 | 161 | 164 | 172
Liters | 0.206 (0.0167) | 0.276 (0.0168) | 0.282 (0.0167) | 0.180 (0.0165)

3. Other Pre Specified Outcome: Change From Baseline (BL) in the Mean Shortness of Breath With Daily Activities (SOBDA) Score for Week 24
Description: The newly developed SOBDA questionnaire assesses dyspnea or shortness of breath (SOB) with daily activities. The SOBDA questionnaire is made up of 13 items completed by the participant (par.) each evening prior to bedtime, when the par. is instructed to reflect on the current day's activities. The daily score is computed as the mean of the scores on the 13 items (>=7 items must have non-missing responses for this to be calculated). The par. is assigned a weekly mean SOBDA score ranging from 1 to 4 (greater scores indicate more severe breathlessness with daily activities) based on the mean of 7 days of data (>=4 of 7 days must be completed for a weekly mean to be calculated). Change from BL is the mean weekly SOBDA score minus BL. Analysis was performed using MMRM with covariates of treatment, BL (mean score in the week prior to treatment), smoking status, center group, week, week by BL and week by treatment interactions. This MMRM analysis only included Weeks 4, 8, 12, and 24.
Time Frame: Baseline and Week 24
Population: ITT Population. Participants analyzed are those with data available at the presented time point; but, all participants without missing covariate information and with >=1 post-Baseline measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | UMEC 125 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD | TIO18 µg QD
Number analyzed (Participants) | 104 | 114 | 117 | 121
scores on a scale | -0.19 (0.041) | -0.29 (0.040) | -0.33 (0.040) | -0.21 (0.040)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the end of treatment (up to 24 weeks).
Description: On-treatment SAEs and non-serious AEs were reported for members of the ITT Population, comprised of all participants randomized to treatment who received at least one dose of randomized study drug in the Treatment Period.
Arm/Group | UMEC 125 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD | TIO18 µg QD
Serious Adverse Events (participants affected / at risk) | 15/222 | 22/217 | 15/215 | 9/215
Other Adverse Events (participants affected / at risk) | 75/222 | 63/217 | 66/215 | 62/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC 125 µg QD (N=222) | UMEC/VI 62.5/25 µg QD (N=217) | UMEC/VI 125/25 µg QD (N=215) | TIO18 µg QD (N=215)
Pneumonia (Infections and infestations) | 2 | 2 | 3 | 2
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 0 | 2 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 6 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal epidural haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC 125 µg QD (N=222) | UMEC/VI 62.5/25 µg QD (N=217) | UMEC/VI 125/25 µg QD (N=215) | TIO18 µg QD (N=215)
Nasopharyngitis (Infections and infestations) | 6 | 14 | 16 | 17
Upper respiratory tract infection (Infections and infestations) | 17 | 6 | 10 | 14
Lower respiratory tract infection (Infections and infestations) | 1 | 8 | 3 | 2
Headache (Nervous system disorders) | 25 | 21 | 20 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 8 | 6 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 7 | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 5 | 8 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 6 | 3
Hypertension (Vascular disorders) | 9 | 1 | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.